CLINICAL TRIAL: NCT03413098
Title: The Evaluation of a Novel Nasal Mask for the Treatment of Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIA233
Record Dates: First submitted 2018-01-22; First posted 2018-01-29 (Actual); Last update posted 2018-03-22 (Actual); Status verified 2018-01

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Trial nasal Continuous Positive Airway Pressure (CPAP) mask (Experimental): Trial nasal CPAP mask
  Interventions: Device: Nasal CPAP mask

INTERVENTIONS:
Device: Nasal CPAP mask — Investigative Nasal Mask to be used for OSA therapy

SUMMARY:
This investigation is a prospective, non randomized, non blinded study. This investigation is designed to evaluate the performance, comfort and ease of use with the F&P trial nasal mask amongst Obstructive Sleep Apnea (OSA) patients.

DETAILED DESCRIPTION:
Visit 1 will involve the participants consented in to the trial. Visit 2 will involve the participants being fitted with the F&P trial nasal mask for use in-home.

The participant will then come in to return the mask (Visit Three) and have a final interview, this ensures the maximum time participants will be exposed to the trial mask in home will be 14 ± 4 days from visit two.

The mask will be returned to the Institution at the conclusion of the trial and the participant will return to their previous mask. The Institution will recruit all patients within 1 week of the beginning of the study.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18+ years of age)
* Able to give consent
* Apnea hypopnea Index (AHI)≥ 5 on diagnostic night
* Prescribed PAP for OSA
* Existing nasal mask user

Exclusion Criteria:

* Inability to give consent
* Patients who are in a coma or a decreased level of consciousness
* Anatomical or physiological conditions making automatic positive airway pressure (APAP) therapy inappropriate (e.g. unconsolidated facial structure)
* Commercial drivers who are investigated by New Zealand Transport Agency
* Current diagnosis of carbon dioxide (CO2) retention
* Pregnant or may think they are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2018-03-09 (Actual); Study Completion 2018-03-09 (Actual)

PRIMARY OUTCOMES:
Ease of use | 2 weeks
  Subjective Questionnaire
Acceptability | 2 weeks
  Subjective Questionnaire

SECONDARY OUTCOMES:
Objective leak data | 2 weeks
  Data obtained from participant's device - Objective

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Gunson, Principal Investigator — Sponsor Employee
Locations (2):
- New Zealand (2):
  - Hastings Memorial Hospital, Hastings
  - WellSleep, Wellington